CLINICAL TRIAL: NCT04477148
Title: Comparison of Intubation Success Rates of Metallic Reusable Laryngoscope Blades and Metallic/Plastic Laryngoscope Blades in Morbidly Obese Patients
Brief Title: Comparison of Intubation Success Rates of 3 Different Laryngoscope Blade Types in Morbidly Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turkish Society of Anesthesiology and Reanimation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Uludaguni
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Intubation;Difficult; Morbid Obesity
Keywords: Intubation; obesity; disposable blade
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metallic Reusable(MR) (Active Comparator): Patients in this group were intubated with reusable metallic blades
  Interventions: Device: endotracheal intubation
- Metallic Disposable(MD) (Active Comparator): Patients in this group were intubated with disposable metallic blades
  Interventions: Device: endotracheal intubation
- Plastic Disposable(PD) (Active Comparator): Patients in this group were intubated with disposable plastic blades
  Interventions: Device: endotracheal intubation

INTERVENTIONS:
Device: endotracheal intubation — patients were intubated with 3 different blades

SUMMARY:
Reusable laryngoscope blades, which are the most commonly used devices for airway management, have been reported to be frequently contaminated and a possible source of infection. Although disposable laryngoscope blades are recommended to reduce the risk of infection, there are studies suggesting increased failed intubation attempt rates.

The major cause of anesthesia-related mortality and morbidity is the failure of airway management. The incidence of difficult airway is reported to be 1-4% in normal population while it ranges up to 12-20% in obese patients. Following the introduction of disposable blades and considering the increased rate of failed intubation in obese patients with these devices, the investigators aimed to make a comparison of successful intubation rates of plastic and metallic disposable blades in morbidly obese patients

DETAILED DESCRIPTION:
Successful airway management is the first and most important step of patient safety in anesthesia practice, and most common reason of morbidity and mortality related to anesthesia is failure to provide optimum airway safety.

Intubation helps the anesthesiologist have complete control over airway by keeping airway open, facilitating control over ventilation, reducing the risk of aspiration and providing safe airway during resuscitation, and laryngoscopes are most commonly used tools for this purpose. Laryngoscope are comprised of a handle and a blade (also contains light source) which are mostly reusable. But these parts are easily contaminated during intubation, creating susceptibility to infection. Some studies report that even handles have a chance of 50% to be contaminated with blood. Insufficiently disinfected blades are also a major source of infection. Laryngoscopes contact with non-intact mucous membranes and blood frequently, thus play an important role in cross contamination. Abramson et al. reported that 1/3 of reusable laryngoscope blades are contaminated with bacteria after multiple uses. Concerns about hygiene and risk of infection (including prion infections) caused many health professionals tend towards use of disposable medical devices. Following their introduction, single use laryngoscope blades have been subject to many studies, and many opinions were discussed in different platforms. In studies in which intubation success rates of metallic reusable, metallic disposable and plastic disposable blades were compared, while some have demonstratedd their success rates to be identical, others concluded that plastic disposable blades were ineffective compared to two other.

Laryngoscopy and endotracheal intubation may not be easily performed in every case. Airway management and endotracheal intubation are easier in non-obese patients compared to obese patients. Short and relatively immobile neck, narrow interincisor distance, hypertrophic tonsillae, uvula and adenoids in obese patients makes intubation more difficult in these patients. Additionally, loss of muscle tonus causes tongue to obstruct airway and epiglottis to touch posterior wall of pharynx, thus obstructing airway further.

The investigators couldn't find any study conducted on obese patients evaluating success rates for intubation of metallic reusable, metallic disposable and plastic disposable blades in the literature. In this study, they aimed to compare intubation success rates of metallic reusable, metallic disposable and plastic disposable blades in intubation of obese patients.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patients with 18-60 years age

Exclusion Criteria:

* less than 3 cm of mouth opening
* airway pathology
* restricted head and neck movement
* expected difficult airway
* sore throat
* upper airway infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2015-04-26 (Actual); Study Completion 2015-06-26 (Actual)

PRIMARY OUTCOMES:
comparison success rate of intubation in three different blades | 3 minutes after anesthesia induction
  The investigators compared reusable metal, single-use metal and single-use plastic blades for their effectiveness in laryngoscopy and intubation in morbid obese patients.

IPD SHARING:
Plan to Share IPD: No